CLINICAL TRIAL: NCT04140409
Title: Sandostatin (Octreotide LAR) May Lead to Clinical Improvement Through Receptor Occupation Optimisation A Prospective Interventional Trial of Patients With Neuro-endocrine Tumors With Carcinoid Syndrome Receiving Octreotide LAR
Brief Title: Sandostatin (Octreotide LAR) May Lead to Clinical Improvement Through Receptor Occupation Optimisation
Acronym: SCIROCCO
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Slow recruitment
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCIROCCO
Record Dates: First submitted 2019-10-22; First posted 2019-10-25 (Actual); Last update posted 2019-10-25 (Actual); Status verified 2019-10

CONDITIONS: Neuroendocrine Tumors; Carcinoid Syndrome
Keywords: NET
MeSH Terms: conditions — Neuroendocrine Tumors; Serotonin Syndrome | interventions — Octreotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): All patients will be treated with octreotide LAR intramuscular injections at maximum doses of 60 mg every 4 weeks or a frequency up to 30 mg octreotide LAR each 2 weeks. Change of dose or frequency is left at the discretion of the investigator until symptom control is obtained.
  Interventions: Drug: Sandostatin

INTERVENTIONS:
Drug: Sandostatin — All patients will be treated with octreotide LAR intramuscular injections at maximum doses of 60 mg every 4 weeks or a frequency up to 30 mg octreotide LAR each 2 weeks. Change of dose or frequency is left at the discretion of the investigator until symptom control is obtained.
  Other Names: Octreotide LAR

SUMMARY:
This is a multi-centric prospective interventional study in which patients with a symptomatic GEP-NET will receive octreotide LAR every 2, 3 or 4 weeks. The basal dose and the dose adaptation will be left at the discretion of the investigator depending on the rate of symptom control. Dose increase up to doses of 60 mg octreotide every 4 weeks, or increase of frequency up to 30 mg every 2 weeks can be done to obtain control of carcinoid symptoms, defined by at least a 50% decrease of the mean number of bowel movements per day and the total number of flushes over 7 days AND a maximum frequency of less than 4 bowel movements a day. If only one symptom is present, analysis will be done for that symptom only: refer to table in statistical analysis The concentration of serum octreotide level will be realized with LCMS/MS following the method of Capron & Wallemacq. Each blood sample should be taken 4 times per year just before the next injection of Octreotide LAR.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent GEP NET Ki 67 ≤ 10 %
* Histologically or cytologically confirmed GEP NET
* Appearance of carcinoid syndrome maximum 6 months before the inclusion
* Evaluable or measurable disease (RECIST 1.1) WHO ECOG performance status 0-2
* Positive somatostatin receptor scintigraphy
* >18 years
* Life expectancy of at least 12 weeks

Exclusion Criteria:

* Uncontrolled concurrent disease which prevents the adequate management and follow-up of the NET.
* Previous malignancy in the last past 3 years except malignancies estimated as completely cured.
* Current pregnancy or breast feeding
* Concomitant anti-tumoral treatment, except external beam radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-02-02 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-09-19 (Actual)

PRIMARY OUTCOMES:
Treatment succes vs treatment failure | 2 years
  The primary endpoint is defined as follows:
  * Treatment success: Symptom control is achieved within 2 years of treatment with octreotide LAR. Symptom control is defined as at least a 50% decrease of the mean number of bowel movements per day and the total number of flushes over 7 days AND a maximum frequency of less than 4 bowel movements a day.
  * Treatment failure: No symptom control is achieved within 2 years of treatment with octreotide LAR.
  The response rate will be calculated as the number of patients with treatment success divided by the total number of included patients that received at least one injection of octreotide LAR.

SECONDARY OUTCOMES:
Symptoms | 2 years
  To describe the number of symptoms in correlation to the serum octreotide level, defined by a blood level test of octreotide.
Rate of diarrhea and flushes | 2 years
  To describe the rate of diarrhea and flushing via a patient diary
Impact of increased dose | 2 years
  To describe the impact of increased dose of octreotide LAR on the symptoms: bowel movements and flushing (via patient diary).
Changes in Quality of life | 2 years
  To describe the effect of Octreotide LAR on Quality of Life, based on the change from baseline in the OLO-GINET21 scores
Effect on tumor control | 2 years
  To describe the effect of Octreotide LAR on tumor control according to RECIST 1.1 criteria
  •
Toxicities | 2 years
  To describe the safety of octreotide (CTCAE grades)
Correlation dose/frequency | 2 years
  To describe the correlation between the dose/frequency of octreotide LAR given and the serum octreotide level.

CONTACTS AND LOCATIONS:
Overall Officials: Ivan Borbath, Prof, Principal Investigator — Cliniques Universitaires St-Luc